CLINICAL TRIAL: NCT04104971
Title: Early and Late Complications of Living Related Pediatric Liver Transplantation
Brief Title: Complications of Pediatric Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Najeb Mohamed, principal investigator, Assiut University
Other Study IDs: liver transplantation
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Liver Transplant; Complications
MeSH Terms: interventions — Hematologic Tests; Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * complete blood count and differential count
  * C-reactive protein , CMV and EBV serology, Liver function ,abdominal Us ,hepatitis markers (A,B ,C ) ,Galactomannan for fungal infection, chest x ray and CT chest.
  * Vascular complications by: Doppler showing (graft size and echopattern ,portal vein, pre and post anastomosis, hepatic veins , biliary passages and hepatic artery resistive index ) and abdominal US .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with complications: children who did liver transplantation and develop complications
  Interventions: Diagnostic Test: blood tests , abdominal US and doppler
- without complications: children who did liver transplantation and do not develop complications
  Interventions: Diagnostic Test: blood tests , abdominal US and doppler

INTERVENTIONS:
Diagnostic Test: blood tests , abdominal US and doppler

SUMMARY:
Liver transplant is the treatment of choice in children with end-stage liver failure.liver transplant is indicated when the risk of mortality from the native liver disease outweighs the overall risk of transplantation.The complications occur both immediately post-transplantation and in the long-term. The main complications in the immediate postoperative period are related to the function of the graft (dysfunction and rejection), the surgical technique, infections (bacterial, fungal, and viral),and systemic problems (pulmonary, renal, or neurological) and in the long term, the complications are typically a consequence of the prolonged immunosuppressive therapy.

DETAILED DESCRIPTION:
Liver transplant is the treatment of choice in children with end-stage liver failure. It involves the surgical removal of the entire organ, which is then replaced with a healthy donor liver. Having a healthy liver is essential to longevity because the liver is responsible for nutrient distribution and toxin removal in the body .

Living-donor liver transplantation has been developed to address the disparity between the number candidates for transplant and the reduced number of available organs for liver transplantation.

In general, liver transplant (LT) is indicated when the risk of mortality from the native liver disease outweighs the overall risk of transplantation. Indications for liver transplantation in children include malignant and non-malignant conditions.

The complications occur both immediately post-transplantation and in the long-term. The main complications in the immediate postoperative period are related to the function of the graft (dysfunction and rejection), the surgical technique, infections (bacterial, fungal, and viral),and systemic problems (pulmonary, renal, or neurological) and In the long term, the complications are typically a consequence of the prolonged immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients from (1- 18) years old who were prepared for liver transplantation and followed up at Yassin Abdel Ghaffar charity center for liver disease and research,Cairo,Egypt. from January 2015 to the end of March 2020.

Exclusion Criteria:

* Any patient who did not survive beyond the first post operative day.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children who were prepared for liver transplantation and followed up at Yassin Abdel Ghaffar charity center for liver disease and research,Cairo,Egypt.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
hematological ,vascular and infectious complications | 5 years
  Number of patients have vascular complications Number of patients have pancytopenia Number of patients have bacterial viral or fungal infection any changes in septic screen of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa HI Abu.Faddan, prof, Study Director — Assiut university children hospital
Locations (1):
- Assiut University Children Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting at march 2020
Access Criteria: through finding the research in the site of ClinicalTrials.gov
URL: http://elhomosany2020@yahoo.com

REFERENCES:
- [Result] Reuben A. Long-term management of the liver transplant patient: diabetes, hyperlipidemia, and obesity. Liver Transpl 2001; 7(Suppl 1): S13-21. Bucuvalas, J., Long-term outcomes in pediatric liver transplantation. Liver Transpl, 2009. 15Suppl 2: p. S6-11. Seyfert-Margolis, V. and S. Feng, Tolerance: is it achievable in pediatric solid organ transplantation? Pediatr Clin North Am, 2010. 57(2): p. 523-38, table of contents. Hackl, C., et al., Current developments in pediatric liver transplantation. World J Hepatol, 2015.7(11): p. 1509-20.